CLINICAL TRIAL: NCT03379857
Title: Prevalence of Strokes Secondary to a Reversible Cerebral Vasoconstriction Attributable to Cannabis Consumption in Young Subjects (≤ 45 Years) Hospitalized for an Ischaemic Stroke
Acronym: CANNASTROKE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6640
Record Dates: First submitted 2017-09-29; First posted 2017-12-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Cannabis Use
MeSH Terms: conditions — Stroke | interventions — Magnetic Resonance Spectroscopy; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: Cannabis User
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabis User (Other)
  Interventions: Other: Drug urinal test

INTERVENTIONS:
Other: Drug urinal test — Non Applicable
  Other Names: Magnetic Resonance Imaging; Computerized Tomography Scan; Transcranial Doppler Ultrasound

SUMMARY:
Incidence of strokes has increased these last 20 years in young population. This rise could be linked to alcohol, tobacco or drug use like cannabis. Cannabis has previously been descripted as a potential factor of reversible vasoconstriction. The main objective is to show that an exhaustive assessment of a stroke facing a young person frequently lead to a diagnostic of reversible vasoconstriction due to cannabis use. Evaluation will focus on prevalence of strokes secondary to a reversible vasoconstriction attributable to cannabis in young subjects.

There's a real public healthcare interest in terms of primary and secondary prevention to evaluate the role of cannabis as a risk factor of stroke in young population.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 18 and 45 years old
* Stroke confirmed by medical imaging
* Written informed consent (subject, nearby or emergency procedure)
* Subject affiliate to a local healthcare insurance office
* For female of childbearing potential, an adequate contraceptive measur

Exclusion Criteria:

* Subject with psychiatric disorder, unable to understand the study or cooperate
* Subject under guardianship or forfeiture of liberty
* Pregnant or breastfeeding woman
* Subject in period of exclusion due to another study or still in follow-up of an interventional study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation Cannabis use | 12 months
Reversible vasoconstriction on medical imaging of intracranial arteries at different moment | 12 months.
  medical imaging of intracranial arteries will show new stenoses (topography, number, evolution), and new ischemic or cerebral haemorrhagic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WOLFF, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (6):
- France (6):
  - Chu Jean Minjoz, Besançon
  - Unite Neuro-Vasculaire, Colmar
  - Chu Bocage, Dijon
  - C.H. G. Muller, Mulhouse
  - Hopital Central, Nancy
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No